CLINICAL TRIAL: NCT04290819
Title: Effects of Creatine and Caffeine Co-Supplementation on Muscle Mass and Muscle Performance in Trained Young Adults
Brief Title: Effect of Creatine and Caffeine on Muscle Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 2018-251
Record Dates: First submitted 2020-01-08; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Performance Enhancing Product Use
Keywords: Muscle Endurance; Strength; Hypertrophy; Resistance Training; Creatine; Caffeine
MeSH Terms: conditions — Hypertrophy | interventions — Creatine; Caffeine

STUDY DESIGN:
Intervention Model Description: 4 groups. Comparing each group against one another. Creatine vs. Caffeine vs. Caffeine and Creatine vs. Placebo
Who Masked: Participant, Investigator
Masking Description: Double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resistance Training with Creatine Monohydrate (Experimental): Participants will go through a 6 week resistance training program (unsupervised), at the facility of their choice. They will be given a program to follow with a 2 day on one day rest split routine as follows: Chest and biceps, legs and core, rest, back and triceps, shoulders and core, rest. This cycle will repeat for the 6 week program.
  Interventions: Dietary Supplement: Creatine Monohydrate
- Resistance Training with Caffeine (Experimental): Participants will go through a 6 week resistance training program (unsupervised), at the facility of their choice. They will be given a program to follow with a 2 day on one day rest split routine as follows: Chest and biceps, legs and core, rest, back and triceps, shoulders and core, rest. This cycle will repeat for the 6 week program.
  Interventions: Dietary Supplement: Caffeine
- Resistance Training with Caffeine and Creatine Monohydrate (Experimental): Participants will go through a 6 week resistance training program (unsupervised), at the facility of their choice. They will be given a program to follow with a 2 day on one day rest split routine as follows: Chest and biceps, legs and core, rest, back and triceps, shoulders and core, rest. This cycle will repeat for the 6 week program.
  Interventions: Dietary Supplement: Creatine Monohydrate and Caffeine
- Resistance Training with Placebo (Placebo Comparator): Participants will go through a 6 week resistance training program (unsupervised), at the facility of their choice. They will be given a program to follow with a 2 day on one day rest split routine as follows: Chest and biceps, legs and core, rest, back and triceps, shoulders and core, rest. This cycle will repeat for the 6 week program.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — 0.1g/kg of body weight (pre measured creatine) and 3mg/kg of body weight (pre measured micronized cellulose powder-caffeine placebo) self administered 1 hr prior to working out mixed in water.
  Arms: Resistance Training with Creatine Monohydrate
Dietary Supplement: Creatine Monohydrate and Caffeine — 0.1g/kg body weight (pre measured creatine) and 3mg/kg body weight (pre measured caffeine) self administered 1hr prior to working out mixed in water.
  Arms: Resistance Training with Caffeine and Creatine Monohydrate
Dietary Supplement: Caffeine — 3mg/kg of body weight (pre measured caffeine) and 0.1g/kg of bodyweight (pre measured maltodextrin- creatine placebo) self administered 1 hr prior to working out mixed in water.
  Arms: Resistance Training with Caffeine
Dietary Supplement: Placebo — 0.1g/kg of body weight (pre measured maltodextrin) and 3mg/kg of body weight (pre measured micronized cellulose powder) self administered 1 hr prior to working out mixed in water.
  Arms: Resistance Training with Placebo

SUMMARY:
To determine if creatine and caffeine can be co-supplemented without inhibiting the effects of creatine.

DETAILED DESCRIPTION:
Creatine and caffeine are among the most popular ergogenic aids used by exercising individuals. Creatine supplementation during resistance training has been shown to increase muscle mass and muscle performance (i.e. strength, endurance), possibly by influencing high-energy phosphate metabolism, muscle protein kinetics, and inflammation. Caffeine ingestion has been shown to increase muscle performance, primarily by influencing adenosine receptor activity, muscle protein kinetics, phosphodiesterase, and excitation-coupling. Previous research investigating the combined effects of creatine and caffeine has produced mixed results, with some showing a beneficial effect on short-term anaerobic type activities, while other report no effect. Despite the potential beneficial effects of creatine and caffeine separately, no study has compared the combined effects of creatine and caffeine during resistance training. Therefore, the purpose of this thesis is to determine the effects of creatine and caffeine co-supplementation during resistance training on muscle mass and muscle performance in trained young adults.

The study will be a double-blind, repeated measures design. In order to minimize group differences, participants will be matched according to age and weight and be randomized on a 1:1:1:1 basis to one of four groups: Creatine + Caffeine (CR-CAF; 0.1 g/kg of creatine monohydrate powder + 3 mg/kg of caffeine [micronized powder]); Creatine (CR; 0.1 g/kg of creatine monohydrate powder + 3 mg/kg of caffeine placebo [micronized cellulose powder]), Caffeine (CAF; 3 mg/kg of caffeine + 0.1 g/kg of creatine monohydrate placebo [maltodextrin]) or placebo (PLA; 0.1g/kg creatine monohydrate placebo + 3 mg/kg of caffeine placebo). An individual, blinded to supplement and group allocation, will be responsible for the preparation of study kits. Each study kit will contain the participants supplement for the duration of the study, detailed supplementation instructions, measuring spoons, supplementation compliance log, daily caffeine consumption log and a resistance training log. Supplement powders will be similar in energy content, color, taste, texture, and appearance. The creatine dosage of 0.1 g/kg has previously been shown to be effective for increasing muscle mass and muscle performance. The caffeine dosage of 3 mg/kg has been shown to increase muscle performance. Participants will be instructed to refrain from additional caffeine sources ≥ 3 hour prior to consuming their supplement so that a valid estimate regarding the effects of caffeine supplementation on muscle can be made. On training days, participants will mix their supplement powder in water and consume the solution 60 minutes prior to exercise. Sixty minutes was chosen because this is the approximate time it takes for peak plasma caffeine concentrations to occur after caffeine ingestion and pre-exercise creatine supplementation has a beneficial effect on muscle performance.

Participants will follow the same periodized, resistance training program for 6 weeks. The program will consist of three sets of 6, 8, 10 repetitions to muscle fatigue in order. Resistance training will start on the first day of supplementation and will consist of a split routine involving whole body musculature. Day 1 will involve chest and biceps musculature and include the following exercises in order: machine-based chest press, free weight incline bench press or dumbbell press, free-weight flat dumbbell press, machine-based pec-dec, free-weight standing barbell curl, free-weight alternate arm dumbbell curl and machine-based preacher curl. Day 2 will involve leg and core musculature and include the following exercises in order: free-weight squat, machine-based leg press, machine-based leg extension, machine-based leg curl, machine-based calf raise, and machine-based weighted abdominal crunches. Day 3 will serve as a rest day from training. Day 4 will involve back and triceps musculature and include the following exercises in order: body weight or weight-assisted chin-ups, machine-based seated row, machine-based lat pull-down, free-weight alternate dumb-bell row, free-weight close-grip bench press, machine-based cable triceps bar extension, and machine-based cable triceps rope extension. Day 5 will involve shoulder and core musculature and include the following exercises in order: free-weight dumbbell press, free-weight upright row, free-weight shrugs, free-weight or machine based lateral deltoid flys, free weight or machine-based rear deltoid flys and machine-based weighted abdominal crunches. Day 6 will serve as a rest day from training. This cycle will be repeated for 6 weeks. Participants will maintain training logs to ensure adherence and compliance to the study and to determine total training volume (load x repetitions x sets).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ages 18-39
* Resistance training for minimum of 6 months 3/week.

Exclusion Criteria:

* Creatine supplementation within last 3 months
* Taking medications that affect muscle biology
* Have a disease that affects muscle biology
* Pre existing liver or kidney abnormalities
* Plan to travel for greater then 1 week during the study where you have NO access to fitness facility.
* Fail Par-Q and are unable to receive doctors clearance

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Muscle strength using a standard plate loaded leg press and chest press machine | 6 weeks
  1-Rep max for leg press and chest press.
Hypertrophy | 6 weeks
  Ultrasound of biceps, triceps, quads and hamstrings. Size in cm of each muscle site.
Muscle endurance using a standard plate loaded leg press and chest press machine | 6 weeks
  Reps to fatigue at 50% 1-Rep Max.
Body Composition using a Bod Pod | 6 weeks
  Test used to determine fat mass and lean tissue within a subject. Gives the fat % and the remainder is considered everything else. Since bone and organ wont really change over 6 weeks, all changes are considered to be lean tissue changes.

SECONDARY OUTCOMES:
Fatigue Scale (Generic) | 6 weeks
  Assessed using fatigue scale (1-10) after each workout. The higher the number, the more the participant is fatigued
Rating of perceived exertion (Generic) | 6 weeks
  Modified to encompass entire training day. 1-10 scale as to how hard that particular workout was. The higher the number, the harder the workout felt to the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Darren G Candow, PhD, Principal Investigator — Assoicate Dean of Kinesiology
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
As of now there is no plan to share data of individual participants.

REFERENCES:
- [Background] Trexler ET, Smith-Ryan AE. Creatine and Caffeine: Considerations for Concurrent Supplementation. Int J Sport Nutr Exerc Metab. 2015 Dec;25(6):607-23. doi: 10.1123/ijsnem.2014-0193. PMID 26219105
- [Background] Candow DG, Chilibeck PD. Timing of creatine or protein supplementation and resistance training in the elderly. Appl Physiol Nutr Metab. 2008 Feb;33(1):184-90. doi: 10.1139/H07-139. PMID 18347671
- [Background] Chilibeck PD, Kaviani M, Candow DG, Zello GA. Effect of creatine supplementation during resistance training on lean tissue mass and muscular strength in older adults: a meta-analysis. Open Access J Sports Med. 2017 Nov 2;8:213-226. doi: 10.2147/OAJSM.S123529. eCollection 2017. PMID 29138605
- [Background] Grgic J. Caffeine ingestion enhances Wingate performance: a meta-analysis. Eur J Sport Sci. 2018 Mar;18(2):219-225. doi: 10.1080/17461391.2017.1394371. Epub 2017 Oct 31. PMID 29087785
- [Background] Kreider RB, Kalman DS, Antonio J, Ziegenfuss TN, Wildman R, Collins R, Candow DG, Kleiner SM, Almada AL, Lopez HL. International Society of Sports Nutrition position stand: safety and efficacy of creatine supplementation in exercise, sport, and medicine. J Int Soc Sports Nutr. 2017 Jun 13;14:18. doi: 10.1186/s12970-017-0173-z. eCollection 2017. PMID 28615996
- [Background] Candow DG, Chilibeck PD, Forbes SC. Creatine supplementation and aging musculoskeletal health. Endocrine. 2014 Apr;45(3):354-61. doi: 10.1007/s12020-013-0070-4. Epub 2013 Nov 5. PMID 24190049
- [Background] Graham TE. Caffeine and exercise: metabolism, endurance and performance. Sports Med. 2001;31(11):785-807. doi: 10.2165/00007256-200131110-00002. PMID 11583104
- [Background] Gualano B, Rawson ES, Candow DG, Chilibeck PD. Creatine supplementation in the aging population: effects on skeletal muscle, bone and brain. Amino Acids. 2016 Aug;48(8):1793-805. doi: 10.1007/s00726-016-2239-7. Epub 2016 Apr 23. PMID 27108136

DOCUMENTS (2):
  • Informed Consent Form (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT04290819/ICF_000.pdf
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT04290819/Prot_001.pdf